CLINICAL TRIAL: NCT04282330
Title: Optimising 3D pH-Weighted CEST MRI in Acute Ischaemic Stroke (CEST in Stroke)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEST in Stroke v4 (03.05.18)
Record Dates: First submitted 2020-02-10; First posted 2020-02-24 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CEST imaging performed (Other): CEST imaging will be performed (15 min): Axial 3D volume acquisition at 3.5 mm isotropic voxel size, 20-30 offset frequencies, plus Axial 3D T1w and T2w map at same resolution for use in CEST quantification. A routine stroke MRI protocol will also be performed (10 min): Axial T2w; Axial DWI and ADC (apparent diffusion coefficient) using accelerated multi-band sequence; Axial T2w* or SWI (susceptibility weighted imaging); and dynamic susceptibility contrast-enhanced (DSC) perfusion imaging following contrast agent administration (5 min, provided Radiology Department protocols allow DSC (e.g. no renal impairment)).
  Interventions: Diagnostic Test: 3D CEST imaging

INTERVENTIONS:
Diagnostic Test: 3D CEST imaging — Chemical Exchange Saturation Transfer (CEST) is an emerging MRI technique that can acquire multiple endogenous contrasts to probe cerebral metabolism.

SUMMARY:
CEST in Stroke is an observational magnetic resonance imaging (MRI) study in acute ischaemic stroke patients. Ischaemic stokes are the most common type of stroke and occur when a blood clot blocks the flow of blood and oxygen your brain needs. This can lead to cellular death (infarction) so the quicker a stroke is diagnosed and treated, the better a patient's recovery is likely to be.

The purpose of this study is to determine the technical feasibility of a new MRI technique known as Chemical Exchange Saturation Transfer (CEST) imaging for assessing the extent of potentially salvageable brain tissue (penumbra) around an area of infarction. CEST imaging works by looking at the chemicals in the brain cells. The chemicals may change when cells are affected by stroke. Stroke patients are not normally treated with with clotbusting drugs or clot-retrieving devices if they arrive at hospital many hours after the stroke because treatment may not help and in some cases it may cause more harm than good. However, the new MRI technique could detect those stroke patients who arrive at hospital many hours after the stroke but still have salvageable brain - in these cases it would be helpful to treat these patients and therefore stop those cells from dying.

However, there are several technical issues that need to be addressed before CEST can be adopted as a routine clinical assessment. CEST in Stroke hopes to address these issues by using an alternate MRI sequence capable of acquiring CEST data over a large portion of the brain in approximately in 10 minutes.

The overall aim of study is to determine the feasibility of CEST imaging for assessing the extent of penumbra, in order to determine which patients may benefit from re-perfusion interventions who would otherwise not be eligible. If the study is successful, further research will be implemented to help clinical decision making in stroke patients who present outside of conventional time windows.

DETAILED DESCRIPTION:
CEST in Stroke is an observational magnetic resonance imaging (MRI) study in acute ischaemic stroke patients. Ischaemic stokes are the most common type of stroke and occur when a blood clot blocks the flow of blood and oxygen your brain needs. This can lead to cellular death (infarction) so the quicker a stroke is diagnosed and treated, the better a patient's recovery is likely to be.

The purpose of this study is to determine the technical feasibility of a new MRI technique known as Chemical Exchange Saturation Transfer (CEST) imaging for assessing the extent of potentially salvageable brain tissue (penumbra) around an area of infarction. CEST imaging works by looking at the chemicals in the brain cells. The chemicals may change when cells are affected by stroke. Stroke patients are not normally treated with with clotbusting drugs or clot-retrieving devices if they arrive at hospital many hours after the stroke because treatment may not help and in some cases it may cause more harm than good. However, the new MRI technique could detect those stroke patients who arrive at hospital many hours after the stroke but still have salvageable brain - in these cases it would be helpful to treat these patients and therefore stop those cells from dying.

However, there are several technical issues that need to be addressed before CEST can be adopted as a routine clinical assessment. CEST in Stroke hopes to address these issues by using an alternate MRI sequence capable of acquiring CEST data over a large portion of the brain in approximately in 10 minutes.

The overall aim of study is to determine the feasibility of CEST imaging for assessing the extent of penumbra, in order to determine which patients may benefit from re-perfusion interventions who would otherwise not be eligible. If the study is successful, further research will be implemented to help clinical decision making in stroke patients who present outside of conventional time windows.

Eligible participants (or a consultee) will be approached upon admission in A&E or on the Hyper Acute Stroke Unit within 24 hours of onset. The study will be described in detail and an information sheet provided. After being given sufficient time to consider participation, the participant or their consultee will be asked to complete a consent form. They will be given a copy of the consent form and information sheet for their records.

A one off study visit will then take place. This will entail a 30 minute MRI scan in the King's College Hospital Clinical Research Facility. In addition, a brief neurological assessment (routine examination for all stroke patients) will also be performed and the following information collected: demographics, past medical history and any local laboratory results. The participant's clinical details will be recorded on a case report form (CRF). Any clinical information not provided by the participant will be completed using the patient's medical notes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute anterior circulation ischaemic stroke
* Within 24 hours of symptom onset as defined by time since last known well
* Measurable neurological deficit (i.e. impairment of one or more of the following: language, motor function, cognition, gaze, vision, neglect)
* National Institutes of Health Stroke Scale (NIHSS) score of >= 10
* >= 18 years old
* Written informed consent from patient, legal representative or consultee

Exclusion Criteria:

* Any contraindication to MRI (e.g. cardiac pacemaker)
* Clinical diagnosis of posterior circulation ischaemic stroke
* NIHSS <10
* Evidence of intracranial haemorrhage or significant non-stroke intracranial pathology (including CNS [central nervous system] neoplasm) on CT
* Seizure at onset of symptoms unless CT identifies positive evidence of significant brain ischaemia (e.g. arterial occlusion, early ischaemic change)
* Planned or anticipated intravenous thrombolysis or endovascular re-perfusion strategies
* Pregnancy
* Known allergy to MRI contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Technical feasibility of 3D CEST imaging in acute stroke: Percentage of patients where acquisition of a comprehensive raw CEST dataset can be performed over the human brain | Within 24 hours of ictus
  Percentage of patients where acquisition of a comprehensive raw CEST dataset can be performed over the human brain
Technical feasibility of 3D CEST imaging in acute stroke: Percentage of patients with quantitative maps of different CEST contrasts produced including APT, NOE, and pH-weighted | Within 24 hours of ictus
  Percentage of patients with quantitative maps of different CEST contrasts produced including APT, NOE, and pH-weighted
Technical feasibility of 3D CEST imaging in acute stroke: Signal-to-noise ratio on the CEST contrasts determined: with and without motion | Within 24 hours of ictus
  Signal-to-noise ratio on the CEST contrasts determined: with and without motion

SECONDARY OUTCOMES:
Clinical feasibility: Number of patients recruited per month (determined at completion of study) | Within 24 hours of ictus
  Number of patients recruited per month (determined at completion of study)
Clinical feasibility: Patients tolerating full scan protocol per month | Within 24 hours of ictus
  Number of patients tolerating full scan protocol per month
Dice score of abnormality seen on CEST contrast & routine stroke sequences | Within 24 hours of ictus
  CEST contrast & perfusion imaging (including PWI-DWI mismatch)

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No